CLINICAL TRIAL: NCT00531232
Title: A Phase IIa Open-label, Dose Confirmation Study of Oral Clofarabine in Adult Patients Previously Treated for Myelodysplastic Syndromes (MDS)
Brief Title: A Dose Confirmation Study of Oral Clofarabine for Adult Patients Previously Treated for Myelodysplastic Syndromes (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLOMDS02507
Record Dates: First submitted 2007-09-14; First posted 2007-09-18 (Estimated); Results first posted 2021-11-02 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Myelodysplastic Syndromes; Secondary Acute Myeloid Leukemia (AML)
Keywords: Previously treated MDS; oral clofarabine; Intermediate-1, Intermediate-2 and High Risk MDS; secondary AML (with history of MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Clofarabine 55 mg/day (Experimental): Participants received Clofarabine 55 mg/day orally for 5 consecutive days of each 28-day treatment cycle until disease progression or death, whichever comes first (maximum study duration: up to 4 years).
  Interventions: Drug: Clofarabine
- Clofarabine 35 mg/day (Experimental): Participants received Clofarabine 35 mg/day orally for 5 consecutive days of each 28-day treatment cycle until disease progression or death, whichever comes first (maximum study duration: up to 4 years).
  Interventions: Drug: Clofarabine
- Clofarabine 25 mg/day (Experimental): Participants received Clofarabine 25 mg/day orally for 5 consecutive days of each 28-day treatment cycle until disease progression or death, whichever comes first (maximum study duration: up to 4 years).
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — Pharmaceutical form: Tablet,
  Route of administration: Oral
  Other Names: Clolar

SUMMARY:
There was no well accepted standard of care for participants who failed or were intolerant to any of the currently approved therapies for myelodysplastic syndromes (MDS). In this study, participants were initially assigned to receive 55 or 35 milligrams (mg) of oral clofarabine daily for 5 days. After safety review of the first participants enrolled, the dose was reduced to 25 milligrams per day (mg/day) for up to 8 cycles as long as the participants continued to benefit and in the absence of progressive disease.

ELIGIBILITY:
Inclusion Criteria:

* Had a pathologically confirmed secondary Acute Myeloid Leukemia ([sAML]; following a history of MDS) or MDS with an intermediate-1 (with marrow blasts greater than or equal to [>=] 5%) or intermediate-2 or high risk score as assessed by the International Prognostic Scoring System at study entry. Participants with refractory anemia with excess blasts in transformation recognized by the French-American-British system, and chronic myelomonocytic leukemia were allowed into the study. Pathologic confirmation was the responsibility of the site investigator.
* Had previously treated MDS defined as follows: a) Participants must had at least one, but no more than two, prior treatment regimens [a.) treatment regimen was defined as any drug or drug combination administered for treatment of MDS with the intent of inducing at least hematologic improvement (consistent with International Working Group criteria); Inadequate treatment, due to drug intolerance or other factors, was considered a prior treatment regimen. Hematopoietic growth factors, hydroxyurea, anti-thymocyte globulin, or supportive care measures (e.g., blood transfusions, immunosuppressive agents, antibiotics) were not considered treatment regimens for the purpose of study entry.] b.) One of the treatment regimens had to be either 5-azacytidine or decitabine. If 5-azacytidine or decitabine was given as a treatment regimen more than once, it was considered as 2 different treatment regimens. c.) Participants could not be refractory (i.e., progression of disease, or no evidence of response, while on the treatment) to more than one prior treatment regimen (to be considered refractory to decitabine or 5-azacitidine, participants must have received >= 4 cycles).
* Had documentation of prior transfusion requirements for the preceding 8 weeks (8 weeks prior to first dose of study drug).
* Had Eastern Cooperative Oncology Group performance status 0-2.
* Was able to comply with study procedures and follow-up examinations.
* Had adequate renal and hepatic functions as indicated by predefined laboratory values: a.) Total bilirubin less than or equal to (<=) 1.5 * institutional Upper Limit of Normal (ULN) except for unconjugated hyperbilirubinemia secondary to treatment for MDS or Gilbert's syndrome; and b.) Aspartate aminotransferase and Alanine aminotransferase <= 2.5*ULN; and c.) Serum creatinine <= 1.0 milligrams per deciliter, then the estimated glomerular filtration rate (GFR) had to be greater than (>) 30 mL/min/1.73 m^2 as calculated by the Modification of Diet in Renal Disease equation.
* Was non-fertile or agreed to use birth control during the study through the end of last treatment visit and at least 90 days after.

Exclusion Criteria:

* Had an adjustment of dose and/or schedule of erythropoietin, granulocyte colony stimulating factor or other growth factors within 8 weeks prior to the first dose of oral clofarabine.
* Had any prior therapy for treatment of sAML. Hydroxyurea must not have been received within 24 hours prior to first dose of study drug.
* Had any other chemotherapy or any investigational therapy within four weeks of first dose of study drug.
* Had any prior pelvic radiotherapy.
* Had a prior hematopoietic stem cell transplant for MDS.
* Had not recovered to <= Grade 2 from any drug-related non-hematologic toxicity prior to first dose of the study drug.
* Had an uncontrolled systemic fungal, bacterial, viral, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Had a psychiatric disorder that would interfere with consent, study participation, or follow-up.
* Had any other severe concurrent disease, or had a history of serious organ dysfunction or disease involving the heart, kidney, or liver, in particular: a.) New York Heart Association classification stage II, III, or IV congestive heart failure; b.) Coronary artery disease or arteriosclerotic cardiovascular disease (angina, myocardial infraction) within 3 months of first dose of study drug; c.) Any other primary cardiac disease that, in the opinion of the investigator, increases the risk of ventricular arrhythmia.
* Had any other severe concurrent disease, or had a history of serious organ dysfunction or disease involving the heart had any prior treatment with Clofarabine.
* Had a diagnosis of another malignancy, unless the participants had been disease-free for at least 3 years following the completion of curative intent therapy with the following exceptions: a.) Participants with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease -free duration, were eligible for this study if definitive treatment for the condition had been completed. b.) Participants with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen values were also eligible for this study if hormonal therapy had been initiated or a radical prostatectomy had been performed.
* Had prior positive test for the Human Immunodeficiency Virus.
* Had currently active gastrointestinal disease, or prior surgery that might affect the ability of the participants to absorb oral Clofarabine.
* Participating in other concurrent investigational protocols that were not restricted to data and/or sample collection for participants demographic and/or sample collection for participants demographic and/or disease purposes.
* Had prior treatment with a known nephrotoxic drug within 2 weeks of the first dose of study drug, unless the participants had a calculated GFR >30 at 2 time points no <7 days apart during the 2-week period prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-05-07 (Actual); Primary Completion 2011-05-12 (Actual); Study Completion 2011-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (6):
- United States (6):
  - The University of Chicago, Chicago, Illinois
  - Weill Medical College of Cornell University, New York, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Baylor University Medical Center Blood Marrow Transplantation Research, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 active centers in United States. A total of 38 participants were enrolled between 07 May 2007 and 07 February 2011.
Pre-assignment Details: Participants initially received either 55 or 35 milligrams per day (mg/day) of Clofarabine orally. After a review of the safety data, the dose was lowered to 25 mg/day; and further participants were enrolled at the 25 mg/day dose level.
Period: Overall Study
Arm/Group | Clofarabine 55 mg/Day | Clofarabine 35 mg/Day | Clofarabine 25 mg/Day
Started | 4 | 9 | 25
Treated | 4 | 8 | 24
Completed | 0 | 0 | 0
Not Completed | 4 | 9 | 25
Not completed — Investigator decision | 0 | 0 | 4
Not completed — Participants refused further treatment | 0 | 1 | 2
Not completed — Adverse events (AEs) | 1 | 2 | 2
Not completed — Treatment failure | 1 | 3 | 7
Not completed — Disease recurrence | 0 | 0 | 1
Not completed — Deceased | 2 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Other | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Analysis was performed on full analysis set (FAS) that included all participants who had received at least 1 dose of oral Clofarabine, regardless of participant's compliance with protocol procedures after enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Clofarabine 55 mg/Day | Clofarabine 35 mg/Day | Clofarabine 25 mg/Day | Total
Number analyzed (Participants) | 4 | 8 | 24 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.0 (4.08) | 68.8 (9.30) | 69.9 (8.68) | 69.9 (8.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 13 | 16
  Male | 3 | 6 | 11 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 3 | 3
  White | 4 | 8 | 21 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response
Description: Overall Response: complete remission(CR) or marrow CR or partial remission (PR), or hematologic improvement (HI) in participants with myelodysplastic syndromes (MDS);CR or CR with incomplete count recovery(CRi),or PR in participants with secondary acute myeloid leukemia (sAML). Per International Working Group (IWG) criteria, CR:<= 5% myeloblasts in bone marrow; persistent dysplasia had to be noted; peripheral blood showing hemoglobin (Hgb)>=11g/dL, platelets >=100*10^9/L,neutrophils >=1*10^9/L, blasts 0%. Marrow CR:<=5%myeloblasts in bone marrow and decreased by >=50% over pretreatment; any HI response in peripheral blood. CRi: meeting all criteria for CR except for residual thrombocytopenia (platelet <100*10^9/L) or neutropenia (ANC <1.0*10^9/L). PR: all CR criteria if abnormal before treatment except that marrow blasts should have decreased by >=50% over pretreatment but still >5%. HI: meeting any of the erythroid, platelet, or neutrophil improvement categories for at least 8 weeks.
Time Frame: From date of randomization until disease recurrence or death, whichever occurred first (maximum study duration: up to 4 years)
Population: Analysis was performed on modified Full Analysis Set (mFAS) that included participants assigned to all doses who had received at least 1 dose of clofarabine, excluding participants treated at 55 mg. Data for this outcome measure (OM) was not planned to be collected and analyzed for Clofarabine 55 mg/day arm.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Clofarabine 35 mg/Day | Clofarabine 25 mg/Day
Number analyzed (Participants) | 8 | 24
percentage of participants | 13 [0.00 to 26.75] | 25 [10.58 to 37.77]

2. Secondary Outcome: Duration of Response (DoR)
Description: DoR: time (in months) from 1st documentation of response to date of 1st documentation of disease relapse, progression or death due to any cause, whichever occured first. Response defined as CR, marrow CR, or PR (MDS participants) and CR/CRi (sAML participants). Per IWG criteria, relapse defined as: return to pretreatment bone marrow blast %; decrease of >=50% from maximum remission levels; reduction in Hgb by >=1.5g/dL.CR:<= 5%myeloblasts in bone marrow; persistent dysplasia; peripheral blood showing Hgb>=11g/dL. Marrow CR:<=5%myeloblasts (bone marrow) and decreased by >=50% over pretreatment; any HI response in peripheral blood. CRi:meeting all criteria for CR except for residual thrombocytopenia/neutropenia. PR: all CR criteria if abnormal before treatment except that marrow blasts should have decreased by >=50%. Progression: at least 50% decrease from maximum remission/response in granulocytes/platelets; reduction in Hgb by >=2g/dL; transfusion dependence. Analyzed by Kaplan-Meier.
Time Frame: From first documentation of response to date of documentation of disease relapse, progression or death due to any cause, whichever occurs first (maximum study duration: up to 4 years)
Population: Analysis was performed on subset of participants who had response. Data for this OM was not planned to be collected and analyzed for Clofarabine 55 mg/day arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Clofarabine 35 mg/Day | Clofarabine 25 mg/Day
Number analyzed (Participants) | 1 | 6
months | 12.5 | 3.2 [1.6 to 6.2]

3. Secondary Outcome: Number of Participants Who Achieved Hematologic Improvement (HI)
Description: Per IWG criteria, HI was defined as meeting any of the erythroid, platelet,and/or neutrophil independence categories for at least 8 consecutive weeks. Erythroid response (pre-treatment,<11 grams per deciliter [g/dL]) was defined as Hgb increased by >=1.5 g/dL;relevant reduction of units of red blood cell (RBC) transfusion by an absolute number of at least 4 RBC transfusion/8 weeks compared with the pretreatment transfusion number in the previous 8 weeks; only RBC transfusions given for Hgb of <=9.0 g/dL pre-treatment counted in the RBC transfusion response evaluation. Platelet response(pretreatment, <100*109/L) was defined as absolute increase of >=30*109/L for participants starting with >20*109/L platelets, increase from <20*109/L to >20*109/L and by at least 100%. Neutrophil response (pre-treatment, <1.0*109/L) was defined by at least 100% increase and an absolute increase >0.5*109/L. Number of participants who achieved HI for MDS participants only was reported in outcome measure.
Time Frame: as for outcome 1
Population: Analysis was performed on mFAS. Data for this OM was not planned to be collected and analyzed for Clofarabine 55 mg/day arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Clofarabine 35 mg/Day | Clofarabine 25 mg/Day
Number analyzed (Participants) | 8 | 24
Participants | 0 | 3

4. Secondary Outcome: Percentage of Participants Achieving Overall Remission (OR)
Description: OR was defined as a best response of CR, marrow CR, or PR in participants with MDS or a best response of CR or CRi in participants with sAML. As per IWG criteria, CR was defined as the following: bone marrow <=5% myeloblasts with normal maturation of all cell lines; persistent dysplasia had to be noted; peripheral blood showing hemoglobin >=11 g/dL, platelets >=100*10^9/L, neutrophils >=1*10^9/L, blasts 0%. Marrow CR was defined as: bone marrow <=5% myeloblasts and decreased by >=50% over pretreatment; any HI response in peripheral blood had to be noted. CRi was defined as meeting all criteria for CR except for residual thrombocytopenia (platelet count <100*10^9/L) or neutropenia (ANC <1.0*10^9/L). PR was defined as all CR criteria if abnormal before treatment except that marrow blasts should have decreased by >=50% over pre-treatment but still >5%. HI was defined as meeting any of the erythroid, platelet, or neutrophil improvement categories for at least 8 weeks.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Clofarabine 35 mg/Day | Clofarabine 25 mg/Day
Number analyzed (Participants) | 8 | 24
percentage of participants | 13 [0.00 to 26.75] | 25 [10.58 to 37.77]

5. Secondary Outcome: Time to Acute Myeloid Leukemia (AML) Transformation
Description: Time to AML transformation was defined as time (in months) from date of the first dose of oral Clofarabine to the date of AML transformation, (i.e., the earliest date when participants experienced bone marrow or peripheral blasts >30%). The analysis was performed by Kaplan-Meier method.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Clofarabine 35 mg/Day | Clofarabine 25 mg/Day
Number analyzed (Participants) | 8 | 24
months | 4.2 [3.1 to NA] — Upper limit of Confidence Interval (CI) was not estimable because the curve's upper CI bound had not crossed 50% survival threshold. | NA [5.2 to NA] — Median was not estimable because the curve's had not crossed 50% survival threshold and upper limit of CI was not estimable because the curve's upper CI bound had not crossed 50% survival threshold.

6. Secondary Outcome: Overall Survival (OS)
Description: OS defined as date of the first dose of oral Clofarabine until date of death due to any cause. If death was not observed, the participant was censored at the earliest of the last date the participant was known to be alive or the study cut-off date. The analysis was performed by Kaplan-Meier method.
Time Frame: From date of first dose of study drug until date of death due to any cause (maximum study duration: up to 4 years)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Clofarabine 35 mg/Day | Clofarabine 25 mg/Day
Number analyzed (Participants) | 8 | 24
months | 4.8 [0.6 to 7.4] | 7.3 [2.8 to NA] — Upper limit of CI was not estimable because the curve's upper CI bound had not crossed 50% survival threshold.

7. Secondary Outcome: Maximum Tolerated Dose (MTD) of Oral Clofarabine
Description: The MTD was the highest dose level of Clofarabine that caused less than (<) 2 participants to experience unacceptable drug-related toxicities after receiving 1 or more of the initial 5 daily doses of Clofarabine. Unacceptable drug-related toxicities included: drug-related prolonged myelosuppression, which was defined as hypocellular bone marrow with <5 percent (%) cellularity at 6 weeks after starting treatment, which required a 1-dose level reduction for subsequent cycles; Common Terminology Criteria for Adverse Events (CTCAE) Grade 4 drug-related non-hematologic toxicity; CTCAE Grade 3 drug-related non-hematologic toxicity that either recovered to Baseline grade but was recurrent to Grade 3 upon re-treatment during the first cycle or did not recover to Grade 1 or Baseline within 3 weeks when the drug was held or dose reduced; drug-related non-hematologic toxicity that resulted in non-completion of at least 4 daily doses of oral Clofarabine at the original assigned dose level.
Time Frame: Cycle 1 (28 days)
Population: Analysis was performed on all participants who received study drug.
Measure: Number; unit: mg/day
Arm/Group | Clofarabine 55 mg/Day | Clofarabine 35 mg/Day | Clofarabine 25 mg/Day
Number analyzed (Participants) | 4 | 8 | 24
mg/day | 25 | 25 | 25

8. Secondary Outcome: Number of Participants With Febrile Neutropenia
Description: Febrile neutropenia was defined as fever (e.g., greater than or equal to (>=) 38.5 Celsius (°C) on a single occasion, or greater than (>) 38°C on 2 occasions within 12 hours) in the setting of neutropenia (defined as Absolute Neutrophil Count <1.0*10^9/liter [L]).
Time Frame: From Baseline up to 45 days post last dose of study drug (maximum study duration: up to 4 years)
Population: Analysis was performed on FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Clofarabine 55 mg/Day | Clofarabine 35 mg/Day | Clofarabine 25 mg/Day
Number analyzed (Participants) | 4 | 8 | 24
Participants | 1 | 1 | 13

9. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Adverse Event (AE): any undesirable physical, psychological/behavioral effect experienced by participant during their participation in clinical study, with study drug usage, whether or not product related.Treatment Emergent AEs (TEAEs): AEs that developed, worsened, or became serious during treatment period (from signature of informed consent form up to 45 days post last dose). Serious AE (SAE):any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization/prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, medically important event. Per National Cancer Institute (NCI)-CTCAE v3.0 severity for each AE were graded as: Grade 1=Mild AE; Grade 2=Moderate AE; Grade 3=Severe AE, Grade 4=Life-threatening/disabling AE and Grade 5=Death related to AE. Participants with TEAEs, SAEs, death, discontinuations, Grade 4 and 5 toxicities were reported.
Time Frame: From Baseline up to 45 days post last dose of study drug (maximum duration: up to 4 years)
Population: Analysis was performed on FAS.
Measure: Count of Participants; unit: Participants
Groups:
- Clofarabine 25 mg/Day: Participants received Clofarabine 25 mg/day orally for 5 consecutive days of each 28-day treatment until disease progression or death, whichever comes first (maximum study duration: up to 4 years).
Arm/Group | Clofarabine 55 mg/Day | Clofarabine 35 mg/Day | Clofarabine 25 mg/Day
Number analyzed (Participants) | 4 | 8 | 24
Participants
  Any TEAE | 4 | 8 | 24
  Any treatment emergent SAE | 4 | 6 | 19
  Any TEAE leading to discontinuation | 1 | 2 | 2
  Any TEAE leading to death | 4 | 7 | 14
  Deaths within 45 days of last dose | 3 | 3 | 3
  Grade 4 Toxicities | 1 | 4 | 18
  Grade 5 Toxicities | 3 | 4 | 4

10. Secondary Outcome: Number of Participants Who Reported Death Within 30 Days of First Dose
Time Frame: Within 30 days of first dose administered on Day 1 of Cycle 1
Population: Analysis was performed on FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Clofarabine 55 mg/Day | Clofarabine 35 mg/Day | Clofarabine 25 mg/Day
Number analyzed (Participants) | 4 | 8 | 24
Participants | 2 | 1 | 1

11. Secondary Outcome: Number of Participants With Unacceptable Drug-related Toxicities During Cycle 1
Description: Unacceptable drug-related toxicities included: drug-related prolonged myelosuppression, which was defined as hypocellular bone marrow with <5% cellularity at 6 weeks after starting treatment, which required a 1-dose level reduction for subsequent cycles; CTCAE Grade 4 drug-related non-hematologic toxicity; CTCAE Grade 3 drug-related non-hematologic toxicity that either recovered to Baseline grade but was recurrent to Grade 3 upon re-treatment during the first cycle or did not recover to Grade 1 or Baseline within 3 weeks when the drug was held or dose reduced; drug-related non-hematologic toxicity that resulted in non-completion of at least 4 daily doses of oral clofarabine at the original assigned dose level. Participants with unacceptable drug-related toxicities during Cycle 1 only was reported in the outcome measure.
Time Frame: Cycle 1 (28 days)
Population: Analysis was performed on FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Clofarabine 55 mg/Day | Clofarabine 35 mg/Day | Clofarabine 25 mg/Day
Number analyzed (Participants) | 4 | 8 | 24
Participants
  Any unacceptable drug-related toxicities | 0 | 1 | 0
  Drug-related prolonged myelosuppression | 0 | 0 | 0
  Grade 4 drug-related non-haematologic toxicity | 0 | 1 | 0
  Grade 3 drug-related recurrent or persistent non-haematologic toxicity | 0 | 0 | 0
  Drug-related toxicity precluding completion of at least 4 daily doses | 0 | 0 | 0

12. Secondary Outcome: Pharmacokinetics (PK) Parameter: Maximum Observed Plasma Concentration (Cmax) of Clofarabine
Description: Cmax was defined as maximum observed plasma concentration of study drug.
Time Frame: Pre-dose and at 1, 3, and 5 hours Post-dose on Day 1 of Cycle 1
Population: Analysis was performed on PK population that included all participants who had received at least 1 dose of oral Clofarabine and had at least 1 sample available for PK analysis.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Clofarabine 55 mg/Day | Clofarabine 35 mg/Day | Clofarabine 25 mg/Day
Number analyzed (Participants) | 4 | 8 | 23
nanograms per milliliter | 158.25 (55.446) | 79.613 (39.597) | 47.813 (44.745)

13. Secondary Outcome: PK Parameter: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Clofarabine
Description: Tmax was defined as the time to reach Cmax (maximum observed plasma concentration).
Time Frame: Pre-dose and at 1, 3, and 5 hours Post-dose on Day 1 of Cycle 1
Population: Analysis was performed on PK population.
Measure: Median (Full Range); unit: hours
Arm/Group | Clofarabine 55 mg/Day | Clofarabine 35 mg/Day | Clofarabine 25 mg/Day
Number analyzed (Participants) | 4 | 8 | 23
hours | 2.02 [1 to 3.03] | 1 [1 to 3] | 2 [0.92 to 4]

14. Secondary Outcome: PK Parameter: Area Under the Concentration-time Curve From Time 0 to Time of Last Measurable Plasma Concentration (AUC0-last) of Clofarabine
Description: AUC0-last was defined as area under the concentration-time curve from time 0 to time of last measurable plasma concentration.
Time Frame: Pre-dose and at 1, 3, and 5 hours Post-dose on Day 1 of Cycle 1
Population: Analysis was performed on PK population.
Measure: Mean (Standard Deviation); unit: nanograms*hours per milliliter
Arm/Group | Clofarabine 55 mg/Day | Clofarabine 35 mg/Day | Clofarabine 25 mg/Day
Number analyzed (Participants) | 4 | 8 | 23
nanograms*hours per milliliter | 590.188 (192.187) | 194.084 (150.035) | 144.604 (124.598)

ADVERSE EVENTS:
Time Frame: AE data were collected from signature of the informed consent form up to 45 days post last dose of study drug (maximum study duration: up to 4 years).
Description: Reported AEs and deaths were TEAEs that developed, worsened, or became serious during the treatment period (from signature of the informed consent form up to 45 days post last dose of study drug). Analysis was performed on FAS.
Arm/Group | Clofarabine 25 mg/Day | Clofarabine 35 mg/Day | Clofarabine 55 mg/Day
All-Cause Mortality (participants affected / at risk) | 14/24 | 7/8 | 4/4
Serious Adverse Events (participants affected / at risk) | 19/24 | 6/8 | 4/4
Other Adverse Events (participants affected / at risk) | 24/24 | 8/8 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine 25 mg/Day (N=24) | Clofarabine 35 mg/Day (N=8) | Clofarabine 55 mg/Day (N=4)
Febrile Neutropenia (Blood and lymphatic system disorders) | 11 (12) | 1 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0)
Splenic Infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial Flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (5) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Enterobacter Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes Simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lobar Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mycobacterium Avium Complex Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oesophageal Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 7 (8) | 2 (2) | 1 (1)
Pneumonia Fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia Streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pseudomonal Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sinusitis Fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Streptococcal Sepsis (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Lactate Dehydrogenase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcus Test Positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Failure To Thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Ureteric Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine 25 mg/Day (N=24) | Clofarabine 35 mg/Day (N=8) | Clofarabine 55 mg/Day (N=4)
Anaemia (Blood and lymphatic system disorders) | 17 (84) | 8 (22) | 3 (10)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (2)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (5) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 20 (134) | 6 (30) | 4 (10)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy Mediastinal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (10) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 20 (107) | 6 (33) | 1 (3)
Retroperitoneal Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (82) | 5 (26) | 1 (7)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic Valve Calcification (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic Valve Disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Dilatation Atrial (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dilatation Ventricular (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left Ventricular Hypertrophy (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Lipomatous Hypertrophy Of The Interatrial Septum (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral Valve Incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Pulmonary Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Supraventricular Extrasystoles (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 7 (9) | 0 (0) | 0 (0)
Tricuspid Valve Incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival Haemorrhage (Eye disorders) | 4 (5) | 1 (1) | 0 (0)
Eye Haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Lacrimation Increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal Haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 3 (3) | 3 (4) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 6 (6) | 2 (2) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (10) | 2 (2) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 5 (5) | 4 (7)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Faecal Incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gingival Bleeding (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Ileus Paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lip Dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Lip Haematoma (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Loose Tooth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Mouth Haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 18 (38) | 6 (20) | 3 (4)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Oral Disorder (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Reflux Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Tongue Discolouration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (14) | 5 (11) | 3 (5)
Asthenia (General disorders) | 8 (9) | 1 (1) | 2 (2)
Chills (General disorders) | 10 (11) | 2 (5) | 0 (0)
Fatigue (General disorders) | 8 (10) | 5 (8) | 2 (4)
Feeling Jittery (General disorders) | 0 (0) | 1 (1) | 0 (0)
Generalised Oedema (General disorders) | 0 (0) | 2 (2) | 1 (1)
Malaise (General disorders) | 3 (3) | 0 (0) | 0 (0)
Mucosal Inflammation (General disorders) | 5 (11) | 3 (4) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 2 (2) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 5 (6) | 0 (0) | 3 (5)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (5) | 1 (2) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Gallbladder Disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic Cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 (5) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fungal Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes Virus Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral Candidiasis (Infections and infestations) | 4 (5) | 0 (0) | 0 (0)
Oral Herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Tooth Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Allergic Transfusion Reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Bloody Airway Discharge (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Transfusion Reaction (Injury, poisoning and procedural complications) | 4 (5) | 2 (2) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 8 (21) | 4 (13) | 2 (3)
Aspartate Aminotransferase Increased (Investigations) | 8 (17) | 4 (15) | 2 (3)
Blood Alkaline Phosphatase Increased (Investigations) | 3 (5) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 6 (21) | 3 (16) | 0 (0)
Blood Creatinine Increased (Investigations) | 3 (5) | 2 (9) | 2 (2)
Cardiac Murmur (Investigations) | 2 (2) | 2 (2) | 1 (1)
Ejection Fraction Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram Qt Prolonged (Investigations) | 2 (2) | 1 (1) | 0 (0)
Electrocardiogram St-T Change (Investigations) | 1 (1) | 2 (2) | 0 (0)
Electrocardiogram St-T Segment Abnormal (Investigations) | 1 (1) | 1 (1) | 0 (0)
Occult Blood Positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Qrs Axis Abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Sputum Culture Positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Troponin I Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urinary Casts (Investigations) | 0 (0) | 2 (3) | 0 (0)
Weight Decreased (Investigations) | 6 (8) | 2 (2) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 8 (8) | 3 (3) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Fluid Overload (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (7) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (2) | 1 (3) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (11) | 0 (0) | 1 (7)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 18 (36) | 1 (7) | 3 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 (15) | 1 (2) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (9) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 17 (45) | 0 (0) | 0 (0)
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Arachnoid Cyst (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral Atrophy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral Ischaemia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 8 (17) | 2 (6) | 3 (3)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3)
Confusional State (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Hallucination, Visual (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (2) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Dysuria (Renal and urinary disorders) | 5 (5) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 7 (10) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ketonuria (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 3 (4) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 8 (11) | 4 (4) | 0 (0)
Renal Cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal Cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Paranasal Sinus Mucosal Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 3 (3) | 2 (2)
Pleural Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Blood Blister (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 0 (0)
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 8 (10) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (7) | 0 (0) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2) | 3 (3)
Rash Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Swelling Face (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Aortic Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 2 (3) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 9 (12) | 2 (3) | 2 (2)
Hypotension (Vascular disorders) | 5 (6) | 1 (1) | 2 (2)
Jugular Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular Calcification (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.